CLINICAL TRIAL: NCT05668208
Title: Comparison of the Effects of Extraperitoneal and Transperitoneal Laparoscopic Surgeries on Intracranial Pressure: A Prospective Clinical Study
Brief Title: Do Extraperitoneal Laparoscopic Surgeries Increase Intracranial Pressure?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Eşref Ulutaş, Medical Doctor (MD), Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 22222222
Record Dates: First submitted 2022-12-11; First posted 2022-12-29 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Intracranial Pressure Increase
Keywords: intracranial pressure; laparoscopic; transperitoneally; extraperitoneal
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- extraperitoneal surgery group - TEP inguinal hernia repair (Experimental): The external sheath of the rectus muscle was seen by passing through the skin and subcutaneous tissue with a mini incision made from the umbilicus edge. A 10 mm trocar was placed in the preperitoneal area and CO2 insufflation was performed. The pressure was set to 14 mmHg. Two more 5 mm trocars were inserted between the umbilicus and the sympisis pubis under the laparoscope. The preperitoneal inguinal area was dissected with a laparoscopic dissector and grasper. The hernia sac was released. A 10x15 cm prolene mesh was spread and fixed to cover the femoral, direct and indirect hernia areas. The trocars were removed by evacuating the CO2 gas. The skin was closed and the operation was terminated.
  Interventions: Device: E-CUBE i7 ultrasound system (Alpinion Medical Systems, Seoul, Republic of Korea)
- transperitoneal surgery group - laparoscopic cholecystectomy (Active Comparator): With a mini incision made under the umbilicus, the abdomen was entered with a 10 mm trocar. Pneumoperitoneum was created with CO2 gas. Intra-abdominal pressure was set to 14 mmHg. Under the guidance of the laparoscope, one 10 mm trocar from the subxiphoid area and two more 5 mm trocars from the subcostal area were inserted. The cystic artery and cystic duct were clipped and cut by exposing the Callot triangle. Then the gallbladder was separated from the liver bed and taken out of the abdomen. The CO2 in the abdomen was evacuated and the trocars were removed. The fascia defect and skin were closed and the operation was terminated.
  Interventions: Device: E-CUBE i7 ultrasound system (Alpinion Medical Systems, Seoul, Republic of Korea)

INTERVENTIONS:
Device: E-CUBE i7 ultrasound system (Alpinion Medical Systems, Seoul, Republic of Korea) — ONSD measurement will be made using the E-CUBE i7 ultrasound system.

SUMMARY:
When the literature is examined, it has been reported in many studies that intracranial pressure increases due to laparoscopic procedures performed in the intraperitoneal area. The mechanism of increased intracranial pressure (ICP) associated with insufflation is most likely due to impaired venous drainage of the lumbar venous plexus at increased intra-abdominal pressure. Changes in ICP can be monitored by ultrasonographic measurement of optic nerve sheath diameter (ONSD), which is a generally accepted simple, reliable and non-invasive ICP measurement technique. In meta-analyses conducted on this subject, it has been revealed that ICP elevation during laparoscopy can be observed with a significant increase in ONSD in the early (0 30 minutes) and late (30-120 minutes) periods during carbondioxid (CO2) pneumoperitoneum.

However, the effect of laparoscopic procedures performed in the extraperitoneal area on the central nervous system is not clear. There is not found any study in the literature comparing laparoscopic procedures, especially performed extraperitoneally and transperitoneally, and their effects on intracranial pressure.

The aim of the study compare to laparoscopic cholecystectomy performed in the transperitoneal area and (totally extra-peritoneal) TEP inguinal hernia repair performed in the extraperitoneal area in terms of intracranial pressure relationship.

DETAILED DESCRIPTION:
A total of 60 patients, including 30 patients who underwent laparoscopic cholecystectomy and 30 patients who underwent TEP inguinal hernia repair between December 2022 and January 2023, were included in the study.

Inclusion criteria: 18-70 years old, ASA (American Society of Anesthesiologists) I-II, patients who will undergo laparoscopic cholecystectomy with the diagnosis of symptomatic cholelithiasis or TEP due to inguinal hernia.

Exclusion criteria: patients who were switched to open surgery, glaucoma, corneal disease, eye surgery, cerebrovascular disease, any neurological disease, chronic kidney disease, liver cirrhosis, and patients whose peritoneum was opened during TEP.

Anesthesia

All patients will undergo general anesthesia and will be given Propofol 2 mg/kg and Fentanyl 2 μg/kg intravenously (IV) for analgesia. Endotracheal intubation will be performed after a 4-minute injection of 0.1 mg/kg Vecuronium. Anesthesia will be maintained with an oxygen-air ratio of 50:50 propofol. For postoperative nausea and vomiting prophylaxis, 4 mg of dexamethasone will be given at induction. Intermittent doses of Fentanyl and Vecuronium will be given from time to time as needed. At the end of the surgery, the neuromuscular paralysis will be reversed with 0.05 mg/kg Neostigmine and 0.02 mg/kg Glycopyrrolate Injection, and the patient will be extubated.

Surgical Method in Patients Undergoing Laparoscopic Cholecystectomy:

With a mini incision made under the umbilicus, the abdomen will be entered with a 10 mm trocar. Pneumoperitoneum will be created with CO2 gas. The intra-abdominal pressure will be set to 14 mmHg. Under the guidance of the laparoscope, 1 10 mm trocar from the subxiphoid region and 2 more 5 mm trocars from the subcostal region will be inserted. The cystic artery and cystic duct will be clipped and cut, exposing the Callot's triangle. The gallbladder will then be separated from the liver bed and removed through the abdomen. The CO2 in the abdomen will be evacuated and the trocars will be removed. The operation will be terminated by closing the fascia defect and the skin.

Surgical Method in Patients with Totally Extra-peritoneal (TEP) Repair:

The outer sheath of the rectus muscle will be seen by passing through the skin and subcutaneous tissue with a mini incision made from the umbilicus. A 10 mm trocar will be placed in the preperitoneal space and CO2 insufflation will be applied. The pressure will be set to 14 mmHg. Two more 5 mm trocars will be placed between the umbilicus and the sympisis pubis under the laparoscope. The preperitoneal inguinal region will be dissected with a laparoscopic dissector and holder. The hernial sac will be released. A 10x15 cm prolene mesh will be fixed to cover the femoral, direct and indirect hernia areas. The trocars will be removed by evacuating the CO2 gas. The skin will be closed and the operation will be terminated.

Results

The primary outcome of the study is the comparison of ONSD measurements between patients who underwent laparoscopic cholecystectomy and TEP repair.

Secondary outcomes are age, gender, ASA score, height, weight, comorbidities, heart rate, blood pressure, oxygen saturation (SpO2), end tidal CO2 (ETCO2) measurements.

ONSD measurement:

ONSD will be performed with transorbital sonography by 2 investigators unaware of the study protocol. Transorbital sonography will be performed using an E-CUBE i7 ultrasound system (mechanical index, 0.2; thermal index, 0) using a linear 6-13 Hz probe (Alpinion Medical Systems, Seoul, Republic of Korea). To prevent eye damage, a sterile occlusion gel will be used and gently probed without applying pressure to the eyelid. Ultrasonographic images of the area will be obtained at the optic nerve level and the ONSD image will be taken 3 mm behind the optic nerve head. The optic nerve sheath will be taken from both eyes at certain times, preoperatively (T0), at the end of insufflation (T1), and at the end of the operation (T2). The average value of the 3 measurements will be recorded as ONSD. Heart rate (HR), blood pressure, SPO2 and EtCO2 will be recorded separately at each time point.

Statistical analysis The primary aim of this study is to compare the effect of laparoscopic surgeries performed in the preperitoneal and intraperitoneal areas on OSD. For clinically reliable results, at least 30 subjects in each group had to detect a difference of 0.3 mm in ONSD measurements. Sample size was calculated based on a pilot study. Multivariate observational analyzes of all data will be performed. Descriptive statistics will be given for hidden variables. Mean and standard deviation will be given for continuous variables, frequency and percentage will be given for categorical variables. Mixed effects models will be created for constant variables. Group, time and group-time interaction will be evaluated. The t-test will be used to measure continuous variables between the 2 groups. When group-time interaction is important, least squares means will be compared. Statistical Analysis SAS (University Edition 9.4) software will be used for data analysis. A P value of <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old,
* ASA (American Society of Anesthesiologists) I-II,
* patients who will undergo laparoscopic cholecystectomy with the diagnosis of symptomatic cholelithiasis or TEP due to inguinal hernia.

Exclusion Criteria:

* patients who were switched to open surgery,
* glaucoma, corneal disease, eye surgery,
* cerebrovascular disease,
* any neurological disease,
* chronic kidney disease,
* liver cirrhosis,
* patients whose peritoneum was opened during TEP.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
measurements of optic nerve sheath diameter (ONSD) | during surgery
  mm

SECONDARY OUTCOMES:
heart rate value | during surgery
  /min
blood pressure | during surgery
  mmHg
SPO2 measurements | during surgery
ETCO2 measurements | during surgery
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Steiner CA, Karaca Z, Moore BJ, Imshaug MC, Pickens G. Surgeries in Hospital-Based Ambulatory Surgery and Hospital Inpatient Settings, 2014. 2017 May [updated 2020 Jul 20]. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #223. Available from http://www.ncbi.nlm.nih.gov/books/NBK442035/ PMID 28722845
- [Background] Montorfano L, Giambartolomei G, Funes DR, Lo Menzo E, Dip F, White KP, Rosenthal RJ. The Cushing reflex and the vasopressin-mediated hemodynamic response to increased intracranial pressure during acute elevations in intraabdominal pressure. Surgery. 2020 Feb;167(2):478-483. doi: 10.1016/j.surg.2019.10.006. Epub 2019 Dec 6. PMID 31813477
- [Background] Rosenthal RJ, Friedman RL, Chidambaram A, Khan AM, Martz J, Shi Q, Nussbaum M. Effects of hyperventilation and hypoventilation on PaCO2 and intracranial pressure during acute elevations of intraabdominal pressure with CO2 pneumoperitoneum: large animal observations. J Am Coll Surg. 1998 Jul;187(1):32-8. doi: 10.1016/s1072-7515(98)00126-4. PMID 9660022
- [Background] Yashwashi T, Kaman L, Kajal K, Dahiya D, Gupta A, Meena SC, Singh K, Reddy A. Effects of low- and high-pressure carbon dioxide pneumoperitoneum on intracranial pressure during laparoscopic cholecystectomy. Surg Endosc. 2020 Oct;34(10):4369-4373. doi: 10.1007/s00464-019-07207-w. Epub 2019 Oct 15. PMID 31617096
- [Background] Robba C, Cardim D, Donnelly J, Bertuccio A, Bacigaluppi S, Bragazzi N, Cabella B, Liu X, Matta B, Lattuada M, Czosnyka M. Effects of pneumoperitoneum and Trendelenburg position on intracranial pressure assessed using different non-invasive methods. Br J Anaesth. 2016 Dec;117(6):783-791. doi: 10.1093/bja/aew356. PMID 27956677
- [Background] Kalmar AF, Foubert L, Hendrickx JF, Mottrie A, Absalom A, Mortier EP, Struys MM. Influence of steep Trendelenburg position and CO(2) pneumoperitoneum on cardiovascular, cerebrovascular, and respiratory homeostasis during robotic prostatectomy. Br J Anaesth. 2010 Apr;104(4):433-9. doi: 10.1093/bja/aeq018. Epub 2010 Feb 18. PMID 20167583
- [Background] Citerio G, Vascotto E, Villa F, Celotti S, Pesenti A. Induced abdominal compartment syndrome increases intracranial pressure in neurotrauma patients: a prospective study. Crit Care Med. 2001 Jul;29(7):1466-71. doi: 10.1097/00003246-200107000-00027. PMID 11445709
- [Background] Rosenthal RJ, Hiatt JR, Phillips EH, Hewitt W, Demetriou AA, Grode M. Intracranial pressure. Effects of pneumoperitoneum in a large-animal model. Surg Endosc. 1997 Apr;11(4):376-80. doi: 10.1007/s004649900367. PMID 9094281
- [Background] Dip F, Nguyen D, Rosales A, Sasson M, Lo Menzo E, Szomstein S, Rosenthal R. Impact of controlled intraabdominal pressure on the optic nerve sheath diameter during laparoscopic procedures. Surg Endosc. 2016 Jan;30(1):44-9. doi: 10.1007/s00464-015-4159-0. Epub 2015 Apr 22. PMID 25899811